CLINICAL TRIAL: NCT06995144
Title: A Randomized, Two-Period, Two-Arm, Double-Dummy, Crossover Study to Compare Natriuretic Effects of Extended Release Torsemide to Immediate Release Torsemide in Patients With Heart Failure (NEXT-HF)
Brief Title: Comparing Natriuretic Effects of ER Torsemide to IR Torsemide in Patients With Heart Failure
Acronym: NEXT-HF
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Sarfez Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SAR-2025-019
Record Dates: First submitted 2025-05-16; First posted 2025-05-29 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Heart Failure; Edema; Pulmonary Congestion; Fluid Overload
Keywords: heart failure; natriuretic; torsemide; Soaanz; extended release; diuretic; sodium retention; water retention; renal clearance; low-sodium; diet; prolonged diuretic action; loop diuretic; urinary sodium excretion; furosemide; bumetanide; chronic kidney disease
MeSH Terms: conditions — Heart Failure; Edema; Hypernatremia; Renal Insufficiency, Chronic

STUDY DESIGN:
Intervention Model Description: Randomized, Two-Period, Two-Arm, Double-Dummy, Crossover Study to Compare Natriuretic Effects of Extended Release Torsemide to Immediate Release Torsemide in Patients with Heart Failure (NEXT-HF)
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm 1 IR torsemide (Active Comparator): Approximately half of the participants will receive 20 mg IR torsemide followed by 24 mg ER torsemide or 40mg IR torsemide followed by 48 mg ER torsemide (6-10 days each)
  Interventions: Drug: Extended Release Torsemide Tablets; Drug: Immedate Release Torsemide Tablets
- ARM 2 ER torsemide (Active Comparator): The other half will receive 24 mg ER torsemide followed by 20 mg IR torsemide, or 48 mg ER torsemide followed by 40 mg IR torsemide (6-10 days each)
  Interventions: Drug: Extended Release Torsemide Tablets; Drug: Immedate Release Torsemide Tablets

INTERVENTIONS:
Drug: Extended Release Torsemide Tablets — Extended release torsemide vs Immediate release torsemide
  Other Names: ER Torsemide tablets
Drug: Immedate Release Torsemide Tablets — Immediate release torsemide vs Extended release torsemide
  Other Names: IR Torsemide Tablets

SUMMARY:
The primary objective of this study is to learn whether a morning dose of extended-release torsemide enhances renal sodium excretion after lunch (4-8 hours after dosing) compared to immediate-release torsemide.

This is a randomized, double-blind, crossover study in patients with heart failure who are on a stable dose of a loop diuretic. During the study period, participants' current loop diuretics will be replaced with an equivalent dose of either immediate-release or extended-release torsemide.

Following a one-week stabilization period on the assigned torsemide formulation, patients will report to the clinical site for an assessment visit. On the study day, patients will take a single dose of the same torsemide formulation they have been on for the past week, administered after breakfast. Urine samples be collected are:

* 0-4 hours post-dosing (pre-lunch period)
* 4-8 hours post-dosing (post-lunch period)
* 8-24 hours post-dosing (24 hours period) The primary endpoint will be urinary sodium excretion (4-8 hours after dosing). This will be compared between the extended-release arm and the immediate-release arm to assess the efficacy of prolonged diuretic action. In addition, urinary potassium and creatinine excretion and creatinine clearance will be measured in all urine samples as the safety endpoints.

DETAILED DESCRIPTION:
Research Plan

Study Design

This is a double-blind, double-dummy, two-period, two-arm, randomized, crossover study.

Initial Study Procedures

Identification of Participants: Patients with a known history of stable heart failure (HF) for at least one month will be identified through healthcare records at clinical site, heart failure clinic, nephrology clinic, and other relevant clinics.

Additionally, providers likely caring for these patients will be contacted to identify potential participants.

Treatment Arms and Crossover Design

* Arm 1: Approximately half of the participants will receive 20 mg IR torsemide followed by 24 mg ER torsemide or 40mg IR torsemide followed by 48 mg ER torsemide (6-10 days each).
* Arm 2: The other half will receive 24 mg ER torsemide followed by 20 mg IR torsemide, or 48 mg ER torsemide followed by 40 mg IR torsemide (6-10 days each).
* Dose Conversion:

  o Patients on 20-40 mg furosemide will be converted to 20 mg IR torsemide or 24 mg ER torsemide.

  o Patients on 60-80 mg furosemide will be converted to 40 mg torsemide (two 20 mg tablets) or 48 mg ER torsemide (two 24 mg tablets).
  * Patients on 1 mg bumetanide will be converted to 20 mg IR torsemide or 24 mg ER torsemide, while those on 2 mg bumetanide will be converted to 40 mg torsemide or 48 mg ER torsemide.
* Double-Dummy Design: To maintain blinding, participants will also receive placebo corresponding to the medications in their arm, ensuring that participants and investigators remain unaware of their treatment assignment.
* Dietary Instructions: Participants will be instructed to follow a low-sodium diet with a daily intake of approximately 3 grams of sodium throughout the study period.

Test Day Procedures

The test day will occur on the last day of each treatment period, with participants staying at the site for 9-10 hours (no overnight stay). The study staff undertake the following:

* Medication Compliance: Collect study medications for pill count and assess compliance.
* Dosing:

  * A standard breakfast will be served 30 minutes before dosing, and participants will be instructed to complete it within 30 minutes.

After completion of breakfast, participants will receive study medication along with 350 ml +/- 20 ml water.

* Post-dose Sample Collection:

  * Urine samples will be collected at 0-4 hours and 4-8 hours after dosing. For each time point,total volume will be measured, and two 5 ml aliquots will be taken for sodium, potassium, and creatinine measurements. The remaining urine will be stored in a cool place for 48 hours or until laboratory results are sent to the site and reviewed by the PI for any discrepancy.
  * After 4 hours post-breakfast, a lunch containing salt will be served, and participants will complete it within 30 minutes.
  * Participants will be instructed to collect urine for the following 16 hours at home to complete the 24-hour collection, with the urine sample returned to the site for recording of volume and processing.
  * Participants will not be permitted to eat except of the site provide breakfast and lunch, and they will be asked consume all the food (breakfast and lunch; no additional snacks or other food items).
  * Participants will be allowed to consume water, but no flavored drinks or sodas, as they require.
  * Participants will be reminded to empty their bladder completely during the each time point. Bladder emptying time (i.e., passing urine) and urine volume will be recorded.
  * After completion of the 4-8 hours urine collection, participants will be given a urine collection container and will be instructed to collect all the urine passed into the container until 24 hours after the dosing time (site will provide dosing time to the participants).
  * The container will be collected next morning by the site personnel, who will bring the container to site. Upon receiving the container, site staff will measure the volume, take two 5 ml aliquots for sample analysis.

Sample Collection Timepoints

• Urine Samples:

o Post-dose Visit 3 (Test Day of Period 1):Collect urine samples at 0-4 hours, 4-8 hours After Test Day of Period 1: 8-24 hours (measure and record total volume for each).

Visit 4 (test day of Period 2): Collect urine samples at 0-4 hours, 4-8 hours. After Test Day of Period 2: 8-24 hours (measure and record total volume for each).

• Blood Samples:

* Visit 1 (screening): Collect 10-12 ml venous blood for CMP-14 with eGFR testing.
* Visit 3 (Test Day of Period 1): Collect 10-12 ml venous blood for CMP-14 with eGFR.
* Visit 4 (test day of Period 2): Collect 10-12 ml venous blood for CMP-14 with eGFR.

Analytes/Measurements

* Blood Samples:

  * Screening: CMP-14 with eGFR
  * Test day of period 1: CMP-14 with eGFR
  * Test day of period 2: CMP-14 with eGFR
* Urine Samples:

  * Test Day (Post-dose 0-4, 4-8, and 8-24 hours): Urine volume, sodium, potassium, and creatinine.

End of Study Procedures

At the end of the study period, participants will:

* Resume their pre-enrollment diuretic regimen.
* Continue routine follow-up with their physicians for standard care.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18 years or older.
* Informed Consent: Willing and able to sign the informed consent form.
* Stable Chronic HF: A clinical diagnosis of chronic heart failure considered stable by the patient's cardiologist/physician or another experienced clinician for at least one month prior to randomization.
* Current Diuretic Therapy: Receiving an oral dose of 20 mg to 80 mg daily of furosemide, or 10 mg to 40 mg daily dose of torsemide, or 1 mg to 4 mg daily dose of bumetanide, for about 30 days prior to randomization.
* Stable HF Medications: No anticipated changes in HF medications during the study period.
* Female Participants: Premenopausal women of childbearing potential must have a negative pregnancy test prior to study initiation and agree to use effective contraceptive methods throughout the study period.

Exclusion Criteria:

* Other Diuretics: Requirement for a diuretic other than furosemide, bumetanide, or torsemide (except for spironolactone, eplerenone, finerenone, or SGLT2 inhibitors) at randomization or during the study.
* Recent Cardiovascular Events: Myocardial infarction, stroke, transient ischemic attack, acute kidney injury, or acute HF requiring hospitalization within 30 days prior to randomization.
* Severe Lung Disease: Severe or symptomatic lung disease or respiratory symptoms distinct from HF.
* Urinary Issues: History of urinary incontinence, or inability to empty the bladder.
* Uncontrolled Comorbidities: Uncontrolled diabetes mellitus or hypertension.
* Renal Dysfunction: Estimated GFR < 30 ml/min/1.72m².
* Cardiac Conditions: History of flash pulmonary edema or amyloid cardiomyopathy.
* Breastfeeding: Female participants who are breastfeeding.
* Recent Participation in Clinical Trials: Participation in another clinical trial within the last three months prior to randomization.
* Requirements for treatment with a non-steroidal anti-inflammatory drug (except for Aspirin up to 200 mg as PRN daily).
* Serum potassium concentration <3.5 or >5.5 mmol/L.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-05-28 (Actual); Primary Completion 2025-12-30 (Actual); Study Completion 2026-03-15 (Estimated)

PRIMARY OUTCOMES:
Urinary sodium excretion measurement | 4-8 hours (post-lunch period)
  Urinary sodium excretion (mmol) measured after dosing: 4-8 hours (post-lunch period)

SECONDARY OUTCOMES:
Urinary sodium excretion | 0-4 hours (pre-lunch period) and 8-24 hours (post-lunch period)
  The secondary endpoints are urinary sodium excretion (mmol) after dosing:
  1. 0-4 hours (pre-lunch period)
  2. 8-24 hours (post-lunch period)
  3. Safety endpoints include:
     * Creatinine clearance (mmol, 0-4, 4-8, and 8-24 hours after dosing)
     * Urinary potassium excretion (mmol, 0-4, 4-8, and 8-24 hours after dosing)

CONTACTS AND LOCATIONS:
Overall Officials: Salim Shah, PhD, JD, Study Chair — Sarfez Pharmaceuticals, Inc.
Locations (1):
- Future Life Clinical Trials, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided
HIPAA